CLINICAL TRIAL: NCT06583304
Title: Clinical Criteria and Hematological Indices in Pediatrics Diagnosed with Familial Mediterranean Fever : a Single Center Study in Upper Egypt
Brief Title: Hematological Indices in Pediatric Diagnosed with Familial Mediterranean Fever
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Mohamed Ahmed Aboelsaud, 71515,Assiut, Assiut University
Other Study IDs: familial Mediterranean fever
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Familial Mediterranean Fever (FMF )
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To investigate the relationship between the hematological indices and subclinical inflammation in FMF patients during their attack-free period, additionally this study aims to assess the potential of these indices as predictive markers for ongoing inflammation in these patients population at Assuit university hospital of pediatrics.

DETAILED DESCRIPTION:
Familial Mediterranean fever (FMF) is the most common hereditary auto inflammatory disease in the world. FMF is caused by gain of function mutations in the MEFV gene, which encodes a protein called pyrin which has regulatory functions on the innate immune system. [1] Mutations interfere with the function of the pyrin domain, initiating an uninterrupted inflammatory cascade [2] Familial Mediterranean fever affects the populations located on the Mediterranean basin. It is virtually limited to Armenians, Turks, Arabs and nonAshkenazi Jews. However, some cases have been described in European countries, including Italy, France, Spain, Portugal and Greece. [3] The clinical presentation of FMF can be variable, likely depending on its genetic heterogeneity and environmental factors. However, the clinical picture is usually very suggestive of the underlying disease. It is typically characterized by recurrent episodes of fever and systemic inflammation with (pleural and peritoneal) serositis and arthritis. Starting in childhood, patients present shortlasting, self-resolving attacks of fever and abdominal, chest, or joint pain with systemic inflammation. Periodicity is not strict and episodes may occur from once a week up to once every three to four months or more in untreated patients. These events are usually very disabling and in clear contrast with complete well-being in attack-free periods [4]. The diagnosis of FMF based on clinical findings is supported by ethnic origin, family history and genetic testing. Several criteria had been developed for the diagnosis of FMF: the most widely used Tel-Hashomer criteria, Most recently, adult and pediatric rheumatology experts have created a new set of classifcation criteria (Eurofever/PRINTO classifcation criteria) [5].

During FMF attacks, many acute phase reactants such as C-reactive protein (CRP), serum amyloid A, fibrinogen, and erythrocyte sedimentation rate (ESR) increase. It is known that a subclinical inflammation continues in FMF patients during the inter attack period and this increases the risk of developing amyloidosis. [6]. Therefore, the use of additional serum markers to evaluate disease activity may provide beneficial advantages for monitoring and preventing further complications. Systemic inflammation also causes changes in the number and composition of circulating blood cells [7] [8]. Neutrophils, lymphocytes and platelets play major roles in systemic inflammation [9]. Neutrophils and platelets secrete proinflammatory cytokines that augment of more neutrophils and platelets [10]. Microparticles released from activated platelets interact with neutrophils through platelet-like lipoxygenase expression and activation of eicosanoid pathway [11]. The platelet count, mean platelet volume (MPV) are the most important indices of platelet function and activation . MPV, a component of routine complete blood count (CBC) tests, is inversely affected by systemic inflammation. MPV levels were shown to be lower in active inflammatory bowel diseases, rheumatoid arthritis (RA) and ankylosing spondylitis (AS) and increased MPV values were reported after treatment. Additionally, the neutrophil-to-lymphocyte ratio (NLR) and the platelet-to-lymphocyte ratio (PLR), which are easily obtained from differential CBC, have been shown to not only increase in inflammation, but also, be correlated with disease activity and prognosis [12] We discuss the clinical criteria and the association of hematological indices with subclinical inflammation and to evaluate their usability as predictors of ongoing inflammation in FMF patients during their attack-free period

ELIGIBILITY:
Inclusion Criteria:

1. Age at enrollment less than18 years.
2. Both sexes.
3. Diagnosed as familial Mediterranean fever according to Tel-Hashomer criteria in pediatrics and Eurofever /PRINTO criteria

Exclusion Criteria:

1- Patients with acute or chronic active infections. 2- Patients with pre-existing illness as chronic lung, liver or renal diseases. 3- Patients with diabetes mellitus, atherosclerotic vascular disease. 4- Patients with malignancy

-

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Their clinical presentation and laboratory finding should fulfill the diagnostic criteria as mentioned by Tel Hashomer criteria in pediatrics (≥2 criteria) and Eurofever /PRINTO criteria (≥6 criteria) and confirmed by genetic testing of the most common 12 genetic variants in MEFV gene
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2024-10-13 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
investigate the association of haematological indices with subclinical inflammation | Baseline
  investigate the association of hematological indices with subclinical inflammation and to evaluate their usability as predictors of ongoing inflammation in FMF patients during their attack-free period in Assiut university hospital and to describe the clinical characteristics of patients diagnosed as FMF in Upper Egypt, and to find the most common presenting symptoms.

REFERENCES:
- [Background] Lancieri M, Bustaffa M, Palmeri S, Prigione I, Penco F, Papa R, Volpi S, Caorsi R, Gattorno M. An Update on Familial Mediterranean Fever. Int J Mol Sci. 2023 May 31;24(11):9584. doi: 10.3390/ijms24119584. PMID 37298536
- [Background] Assouad E, El Hage S, Safi S, El Kareh A, Mokled E, Salameh P. Familial Mediterranean fever research activity in the Arab world: the need for regional and international collaborations. East Mediterr Health J. 2021 Oct 27;27(10):984-992. doi: 10.26719/emhj.21.036. PMID 34766324
- [Background] Tufan A, Lachmann HJ. Familial Mediterranean fever, from pathogenesis to treatment: a contemporary review. Turk J Med Sci. 2020 Nov 3;50(SI-2):1591-1610. doi: 10.3906/sag-2008-11. PMID 32806879